CLINICAL TRIAL: NCT05050565
Title: Psychological Flexibility in Chronic Pain Populations; an Observation- and Validation Study
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: 20210629
Record Dates: First submitted 2021-08-31; First posted 2021-09-20 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Chronic Pain
Keywords: chronic pain; psychological flexibility; stigma
MeSH Terms: conditions — Chronic Pain; Social Stigma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Experiences of stigma and psychological flexibility in chronic pain participants — Chronic pain participants will answer questionnaires at two points in time, two weeks apart. These questionnaires ask about stigma and psychological flexibility, as well as depression, catastrophizing, pain interference, and social adjustment. The data collected is only observational and does not include any intervention.

SUMMARY:
Chronic pain in general is a substantial problem and is a source of a great deal of disability and suffering. It is known that processes like stigma and psychological flexibility (PF) play a significant role in these outcomes. At the same time, there are many specific chronic pain disorders and there is less knowledge about similarities and differences between these specific conditions, whether the role of processes like these vary between conditions or not. For studies that can address this to be done in Sweden, there will need to be adequately translated and validated measures of the key processes identified.

The main aim of the current study is to look at whether the role of PF and stigma in pain-related outcomes differ across pain conditions. In support of that, a secondary aim is to first validate measures of stigma and PF in chronic pain populations. For this secondary aim, the current study seeks to investigate the factor structure, construct - and criterion validity, internal consistency, and test-retest reliability of a Swedish version of the Multidimensional Psychological Flexibility Inventory (MPFI) as well as of a Swedish version of the Stigma Scale for Chronic Illnesses (SSCI-8).

DETAILED DESCRIPTION:
Chronic pain is related to impaired everyday functioning and social adjustment, such as working ability or engaging in recreational activities, and to emotional suffering, such as depression. Sexual functioning and satisfaction may be impaired for patients with vulvodynia and in some cases for patients with endometriosis. Pain seems to interfere with sexual functioning even for people with low back pain and fibromyalgia. Chronic pain is also related to anxiety, and the chronic pain literature often highlights the role of catastrophizing thoughts in exacerbating the experience of pain. Stigma and psychological flexibility (PF) appear to play a role in the suffering endured by people with chronic pain, but it is less clear how these processes differ, or not, between specific pain conditions such as, but not limited to, fibromyalgia, chronic low back pain, endometriosis and vulvodynia. Thus, the main aim of the current study is to investigate this by having participants with various chronic pain conditions fill out measures on stigma and psychological flexibility, and to see how these processes differ across conditions.

However, there is currently a lack of measures in Swedish to adequately capture stigma and psychological flexibility satisfactory. A secondary aim is thus to validate a Swedish version of the Multidimensional Psychological Flexibility Inventory (MPFI) and the Stigma Scale for Chronic Illnesses (SSCI-8).

In order to establish construct- and criterion validity, scores on these measures will be compared to that of related outcomes such as specific facets of psychological flexibility, pain interference, depression, social adjustment, and catastrophizing. In addition, test-retest reliability, internal consistency and factor structures for each measure, the SSCI-8 and the MPFI will be examined.

If eligible, participants will be directed to answer questionnaires via RedCap, a GDPR-compliant mobile application. After finishing the questionnaires, the participants will be reminded after two weeks in order to fill out the same questionnaires once more. At this second time point, questions regarding participant characteristics such as demography and pain background will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or over
* Suffering from chronic or recurrent pain for ≥ 3 months
* Access to an internet enabled phone/computer/tablet
* Fluent in written Swedish
* Willing to be contacted during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People suffering from a chronic pain condition, such as fibromyalgia, chronic back pain, endometriosis, vulvodynia, or other chronic pain conditions.
Sampling Method: Non-Probability Sample
Enrollment: 404 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2022-01-04 (Actual); Study Completion 2022-01-04 (Actual)

PRIMARY OUTCOMES:
Stigma Scale for Chronic Illnesses (SSCI-8) | Measured immediately following participant consent to undertake survey, and again two weeks thereafter
  The SSCI-8 is an eight-item measure including items reflecting both enacted and internalized stigma. Minimum score is 8, and maximum score is 40. Higher scores indicate a greater degree of stigma. It is administered alongside the other outcomes in order to establish validity. It is also administered in order to examine similarities and dissimilarities between different chronic pain conditions in the stigma experience and in its relationship to the other outcome measures. The SSCI-8 will be administered a second time in order to examine temporal stability of the instrument.
Multidimensional Psychological Flexibility Inventory (MPFI) | Measured immediately following participant consent to undertake survey, and again two weeks thereafter
  The MPFI is a 60-item measure reflecting all facets of psychological flexibility. The measure is divided into two overarching dimensions, namely inflexibility and flexibility. Each dimension contains 30 items, and in each dimension the minimum score is an average of 1 across the 30 items, while the maximum score is an average of 6 across the 30 items. For the inflexibility part of the MPFI, a higher average score indicates higher inflexibility. For the flexibility part of the MPFI, a higher average score indicates higher flexibility. The MPFI is administered alongside the other outcomes in order to establish validity. It is also administered in order to examine similarities and dissimilarities between different chronic pain conditions in psychological flexibility and in its relationship to the other outcome measures. The MPFI will be administered a second time in order to examine temporal stability of the instrument.

SECONDARY OUTCOMES:
Chronic Pain Acceptance Questionnaire (CPAQ-8) | Measured immediately following participant consent to undertake survey, and again two weeks thereafter
  An eight-item measure on pain acceptance. The minimum score is 0, and the maximum score is 48. Higher scores indicate higher pain acceptance.
Committed Action Questionnaire 8-item version (CAQ-8) | Measured immediately following participant consent to undertake survey, and again two weeks thereafter
  An eight-item measure on committed action. The minimum score is 0, and the maximum score is 48. Higher scores indicate higher levels of committed action.
Five Facet Mindfulness Questionnaire (FFMQ) - acting with awareness facet | Measured immediately following participant consent to undertake survey, and again two weeks thereafter
  An eight-item subscale on acting with awareness. The minimum score is 8, and the maximum score is 40. It is possible to divide the summary score into an average score. If so, the minimum average score is 1, and the maximum average score is 5. Higher scores indicate lower levels of acting with awareness.
Patient Health Questionnaire (PHQ-9) | Measured immediately following participant consent to undertake survey, and again two weeks thereafter
  A nine-item measure on symptoms of depression, with a minimum score of 0 and a maximum score of 27. Higher scores indicate higher levels of depression. The scale also includes as additional item regarding how the depressive symptoms have interfered with everyday functioning.
Coping Strategy Questionnaire (CSQ) - catastrophizing subscale | Measured immediately following participant consent to undertake survey, and again two weeks thereafter
  A six-item subscale on pain catastrophizing. The minimum score is 0 and maximum score is 36. Higher scores indicate higher levels of catastrophizing.
Work and Social Adjustment Scale (WSAS) | Measured immediately following participant consent to undertake survey, and again two weeks thereafter
  The WSAS is a five-item measure on social adjustment. The minimum score is 0 and maximum score is 40. Higher scores indicate lower work and social adjustment.
Brief Pain inventory - short form (BPI-SF) | Measured immediately following participant consent to undertake survey, and again two weeks thereafter
  For this study, two items on pain severity, one regarding average pain severity during the last week and one regarding pain severity at the current moment, and nine items on pain interference will be used. Two out of the nine pain interference items, exploring how pain interferes with sexual activities and enjoyment of sex, have been created and added by the research team. The two pain severity items are each scored from 0 to 10, with 0 indicating the least amount of pain and 10 indicating the highest amount of pain. The original seven pain interference items are each scored in the same way, but can also together generate an average score, with the minimum average score then being 0 and the maximum average score being 10. A higher score indicates a higher level of pain interference. The two pain interference items created by the research team are each scored from 0 to 10, with 0 indicating the least amount of interference and 10 indicating the highest amount of interference.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Buhrman, PhD, Principal Investigator — Uppsala University
Locations (1):
- Department of Psychology, Uppsala University, Uppsala, Uppland, Sweden

REFERENCES:
- [Derived] Sundstrom FT, Lavefjord A, Buhrman M, McCracken LM. Assessing Psychological Flexibility and Inflexibility in Chronic Pain Using the Multidimensional Psychological Flexibility Inventory (MPFI). J Pain. 2023 May;24(5):770-781. doi: 10.1016/j.jpain.2022.11.010. Epub 2022 Nov 25. PMID 36442815